CLINICAL TRIAL: NCT04134403
Title: Steroids, Thiamine and Ascorbic Acid Supplementation in Septic Shock (STASIS): A Prospective Crossover Randomized Controlled Study
Brief Title: Steroids, Thiamine and Ascorbic Acid in Septic Shock
Acronym: STASIS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Baqiyatallah Medical Sciences University (Other)
Collaborators: Hamadan University of Medical Science (Other); Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir Vahedian-Azimi, Principle Investigator, Associate Professor, Baqiyatallah Medical Sciences University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STASIS
Record Dates: First submitted 2019-09-18; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Septic Shock
Keywords: Steroids; Thiamine; Ascorbic Acid Supplementation; Septic Shock; STASIS
MeSH Terms: conditions — Shock, Septic | interventions — IbsC protein, E coli

STUDY DESIGN:
Intervention Model Description: A Prospective Parallel Randomized Controlled clinical Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Intervention (Experimental): Arm will be those that are randomized to receive usual care plus hydrocortisone, thiamine and ascorbic acid.
  Interventions: Drug: STASIS
- Arm 2: Usual care (No Intervention): Arm will be those that are randomized to receive usual care alone.

INTERVENTIONS:
Drug: STASIS — Hydrocortisone sodium succinate, 50 mg, every 6 hours, 7 days or until ICU discharge Thiamine, 200 mg, every 12 hours, 4 days or until ICU discharge Ascorbic acid, 1,500 mg, every 6 hours, 4 days or until ICU discharge
  Arms: Arm 1: Intervention

SUMMARY:
The objective of this project is to determine if in patients admitted to the hospital with septic shock (population), does treatment with a bundle including hydrocortisone, thiamine, and ascorbic acid improve in-hospital or 28-day mortality (primary outcomes) or surrogate markers of illness severity including: (1) ICU or hospital length-of-stay, (2) duration of invasive mechanical ventilation, (3) duration of vasopressor administration, (4) incidence and severity of ICU delirium, and (5) illness severity (secondary outcomes).

DETAILED DESCRIPTION:
This trial is designed as a multi-center prospective, double-blinded, randomized controlled study. The objective of this project is to determine if in patients admitted to the hospital with septic shock (population), does treatment with a bundle including hydrocortisone, thiamine, and ascorbic acid improve in-hospital or 28-day mortality (primary outcomes) or surrogate markers of illness severity including: (1) ICU or hospital length-of-stay, (2) duration of invasive mechanical ventilation, (3) duration of vasopressor administration, (4) incidence and severity of ICU delirium, and (5) illness severity (secondary outcomes). The calculated sample size is 80. Subjects will be followed for 28 days or until hospital discharge.

Patients eligible for inclusion must be admitted with septic shock (as defined by SEPSIS-3) requiring vasopressors to maintain MAP ≥ 65 AND serum lactate level >2 mmol/L after adequate fluid resuscitation (generally recognized at 30 ml/kg crystalloid unless contraindicated as deemed by treating clinician) within the first three hours.

The exclusion criteria are: age < 18 years, pregnant, patients with limitation of care (i.e. do not resuscitate [DNR]), known Glucose-6-Phosphate Dehydrogenase (G6PD) Deficiency, and vasopressor use for > 24 hours prior to study enrollment.

Patients in Arm 1 will randomized to receive usual care + hydrocortisone, thiamine and ascorbic acid. Arm 2 will be randomized to receive usual care alone. Crossover is not allowed. If a patient is randomized into study Arm 2, the treating physician may decide to administer study medications if they feel it is in the best interest of the patient. In this case the patient will continue to be analyzed in their assigned arm on an intention to treat basis. Source of participants will be in-hospital and Emergency Department patients.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock admitted to the ICU within 24 hours as defined by SEPSIS-3
* SEPSIS-3 defines septic shock as sepsis with the following criteria despite adequate fluid resuscitation:

  * Vasopressor required to maintain MAP ≥ 65 AND
  * Serum lactate level >2.0 mmol/L
* Age ≥ 18 years
* Non-pregnant
* Ability to consent with medical capacity or legally authorized representative (LAR) consent

Exclusion Criteria:

* Age < 18 years
* Pregnant defined by negative serum HCG in all females
* Patients with limitation of care (i.e. DNR)
* Known G6PD deficiency
* Excluding primary admission diagnosis including the following:

  * Acute stroke
  * Acute coronary syndrome
  * Active gastrointestinal bleed
  * Burn
  * Trauma
* Prisoners
* >1 episode of sepsis in hospital admission
* Vasopressor use prior to randomization for more than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
In-hospital or 28-day mortality rate | 28 days or discharge (whichever comes first)
  To determine if the addition of hydrocortisone, thiamine and ascorbic acid to standard care versus standard care in septic shock confers an in-hospital and 28-day mortality benefit

SECONDARY OUTCOMES:
Illness Severity (Change in SOFA Score) | 72 hours
  To determine if the addition of hydrocortisone, thiamine and ascorbic acid to standard care in septic shock confers more rapid improvements in illness severity
Hospital length-of-stay ICU LOS Duration of intubation | 1 year or discharge (whichever comes first)
  To determine if the addition of hydrocortisone, thiamine and ascorbic acid to standard care in septic shock confers improved hospital length-of-stay metrics
ICU length-of-stay | 90 days or discharge (whichever comes first)
  To determine if the addition of hydrocortisone, thiamine and ascorbic acid to standard care in septic shock confers improved ICU length-of-stay metrics
Vasopressor duration (days) | 28 days or discharge (whichever comes first)
  To determine if the addition of hydrocortisone, thiamine and ascorbic acid to standard care in septic shock confers improvement in vasopressor requirements
ICU delerium (CAM-ICU score) | 28 days or discharge (whichever comes first)
  To determine if the addition of hydrocortisone, thiamine and ascorbic acid to standard care in septic shock changes the incidence or severity of ICU delerium
Mechanical ventilation | 28 days or discharge (whichever comes first)
  To determine if the addition of hydrocortisone, thiamine and ascorbic acid to standard care in septic shock changes the incidence or duration of invasive mechanical ventilation.
Cardiac arrest | 28 days or discharge (whichever comes first)
  To determine if the addition of hydrocortisone, thiamine and ascorbic acid to standard care in septic shock changes the incidence of cardiac arrest or need for cardiopulmonary resuscitation
Renal replacement therapy | 28 days or discharge (whichever comes first)
  o determine if the addition of hydrocortisone, thiamine and ascorbic acid to standard care in septic shock changes the incidence of cardiac arrest or need for renal replacement therapy.
C-reactive protein | 28 days or discharge (whichever comes first)
  To determine if the addition of hydrocortisone, thiamine and ascorbic acid to standard care in septic shock changes the biochemical profiling in septic patients including a more rapid improvement in C-reactive protein
Procalcitonin | 28 days or discharge (whichever comes first)
  o determine if the addition of hydrocortisone, thiamine and ascorbic acid to standard care in septic shock changes the biochemical profiling in septic patients including a more rapid improvement in procalcitonin.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Vahedian-Azimi, PhD, Principal Investigator — Baqiyatallah University of Medical Scienecs; Andrew C Miller, MD, Principal Investigator — East Carolina University

IPD SHARING:
Plan to Share IPD: No